CLINICAL TRIAL: NCT07201714
Title: Oral L-Carnitine Supplementation in Cardiorenal Heart Failure Patients
Brief Title: Oral Carnitine in Heart Failure Patients
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Chris McIntyre, Nephrologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 16078
Record Dates: First submitted 2025-06-20; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Carnitine Deficiency
MeSH Terms: conditions — Heart Failure; Systemic carnitine deficiency | interventions — Carnitine

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Oral Levocarnitine (L-Carnitine), 2970mg daily dose (990mg taken 3 times a day) for 3 months.
  Interventions: Drug: Levocarnitine

INTERVENTIONS:
Drug: Levocarnitine — Oral L-carnitine, 2970mg daily (950mg, to be taken 3 times a day) for 3 months.

SUMMARY:
Heart failure is a condition in which the heart is unable to pump blood effectively, leading to symptoms like being more tired, shortness of breath, and swelling in the body. Carnitine is a naturally occurring substance in the body that plays a role in turning fat into energy. This study will determine whether oral L-Carnitine supplementation can improve symptoms, enhance heart function and possibly improve the quality of life in individuals with heart failure.

DETAILED DESCRIPTION:
Heart failure (HF) is a multi-organ syndrome that is fundamentally driven by metabolic failure. Metabolic alterations include reduced fatty acid oxidation, which is the main fuel source for cardiac myocyctes in normal circumstances. Carnitine is a vitamin-like modified amino acid that is essential in the oxidation of fatty acids and has been found to be reduced in the heart failure population. Abnormalities in carnitine metabolism are thought to contribute to myocardial dysfunction, oxidative stress and inflammation. Carnitine supplementation may increase fatty acid oxidation, and therefore energy metabolism in heart failure patients, thus improving functional capacity, clinical measures and quality of life in this vulnerable patient population.

ELIGIBILITY:
Inclusion Criteria:

* Clinical-pathological diagnosis of heart failure with some degree of cardiorenal syndrome
* Stage 1, 2, 3a, 3b, or 4 chronic kidney disease
* Age ≥ 18 years
* Able to speak and read English
* Willing and able to provide consent

Exclusion Criteria:

* Estimated GFR <15 mL/min/1.73m2 or Stage 5 chronic kidney disease
* Currently undergoing renal replacement therapy of any kind
* Pregnant, breastfeeding or intending pregnancy
* History of seizures of any type
* Known allergy to levocarnitine, magnesium stearate, microcrystalline cellulose or povidone
* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | From study start to end of study at 52 weeks
  % of eligible patients enrolled over the study period
Retention Rate | From enrollment to end of treatment at 6 months
  % of enrolled participants completing final follow up
Intervention adherence | From enrollment to end of study treatment at 6 months
  Medication compliance measured by the % of prescribed L-carnitine doses taken. Pill counts will be completed at the end of the medication intervention time period at Visit 2.
Safety and Tolerability (adverse events) | From enrollment to end of treatment at 6 months
  Participants will be monitored throughout the study for any adverse events.
Data Completeness | From start of study to end of study at 52 weeks
  % of participants with complete data for each outcome

SECONDARY OUTCOMES:
Change in Patient Reported Outcome Measurements (PROM) using the Dynamic Patient Reported Outcome Measure (d/PROM) | From enrollment to the end of treatment at 6 months.
  dPROm questionnaire is a digital application patient reported tool which uses a visual analogue scale to measure 3 domains (symptoms, health-related QoL and limitations) using a total of 12 questions. Participants will be assigned a unique unidentifiable username and password and be asked to complete the questionnaire daily over the course of the study.
Change in cognitive function (Montreal Cognitive Assessment (MoCA)) | From enrollment to the end of treatment at 6 months.
  The MoCA test is a validated and highly sensitive tool for the detection of mild cognitive impairment. The MoCA accurately measures short term memory; visuospatial abilities; executive functions; attention, concentration and working memory; language; and orientation to time and place.
Change in cognitive function (Creyos) | From enrollment to the end of treatment at 6 months.
  Creyos is an easily administered validated and engaging cognitive assessment. Creyos uses an online platform to deliver scientifically rigorous neurocognitive tasks and batteries based on classical paradigms from cognitive psychology literature. The tests that are used in Creyos are designed to measure cognition in scientific studies and clinical trials. The brain games presented in Creyos encompass testing to assess short-term memory, reasoning, attention and verbal ability.
Change in Patient Reported Outcome Measurements (PROM) using Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | From enrollment to the end of treatment at 6 months.
  KCCQ-12 is a validated and standardized commonly used PROM in the heart failure population. It consists of 12 questions that map 7 different domains: symptom frequency; symptom burden; symptom stability; physical limitations; social limitations; quality of life; and self-efficacy. Scores are represented on a 0-100-point scale, with lower scores representing more severe symptoms and limitations.
Change in Cardiac Function (Echocardiogram) | From enrollment to the end of treatment at 6 months.
  An echocardiogram will be completed at each visit. Images will be captured in the left lateral position and standard apical 2, 3 and 4 chamber views will be recorded for analysis. Three cardiac cycles will be recorded for each time point and values will be derived for segmental and global longitudinal strain.
Change in Functional Capacity (hand-grip strength (HGS) | From enrollment to the end of treatment at 6 months.
  A Smedley hand grip dynamometer will be used to measure HGS. Participants will be tested in a sitting position with shoulder adducted and neutrally rotated with the elbow flexed at 90o. The participant will be asked to squeeze the handle of the dynamometer as hard as possible for 5 seconds and then relax. The best value out of three attempts will be recorded in kilograms.
Change in Functional Capacity (6-minute walk test) | From enrollment to the end of treatment at 6 months.
  The 6-minute walk test measures functional exercise capacity in an objective way. The test procedure is used when a patient would not be able to perform a cardiopulmonary exercise test. (stress test) due to chronic disease (eg Heart Failure)
Change in Functional Capacity using Sit to Stand Test (STST) | From enrollment to the end of treatment at 6 months
  The sit to stand test has been shown to be a reliable alternative to the 6-minute walk test and may be used in patients who are assessed or who feel that they may not be able to complete a 6-minute walk test due to mobility issues.

OTHER OUTCOMES:
Change in serum biomarkers | From enrolment to the end of treatment at 6 months.
  A blood sample will be collected at each visit to compare any changes in heart failure and inflammatory markers. (Beta-natriuretic protein (BNP), C-reactive protein (CRP), Cytokine levels, cholesterol panel, Lp (a), albumin, total protein, INR, PTT, creatinine, urea, Trimethylamine N-oxide (TMAO)
Change in urine biomarkers | From enrolment to the end of treatment at 6 months.
  A urine sample will be collected at each visit to assess measures of renal and metabolic function. (carnitine, sodium, osmolality, ketone metabolites, myoglobin, TMAO)

CONTACTS AND LOCATIONS:
Overall Officials: Chris McIntyre, MBBS DM, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Not yet determined